CLINICAL TRIAL: NCT06608342
Title: Clinical Study of Autologous Hematopoietic Stem Cell Transplantation Combined With CD19-CART Treatment for Adult High-risk Acute Lymphoblastic Leukemia
Brief Title: Autologous Hematopoietic Stem Cell Transplantation Combined With CD19-CART Treatment of Adult High-risk Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024036
Record Dates: First submitted 2024-09-06; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Acute Lymphoblastic Leukemia ALL
Keywords: inaticabtagene autoleucel; auto-HSCT
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous hematopoietic stem cell transplantation combined with CD19-CART (Experimental)
  Interventions: Biological: Autologous hematopoietic stem cell transplantation combined with CD19-CART

INTERVENTIONS:
Biological: Autologous hematopoietic stem cell transplantation combined with CD19-CART — Autologous CD19-CAR T cells were transfused +7 days after autologous hematopoietic stem cell transplantation

SUMMARY:
To observe the efficacy and side effects of autologous hematopoietic stem cell transplantation combined with CD19-CART for adult acute lymphoblastic leukemia, and to evaluate the safety and efficacy of this regimen in the treatment of acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
To observe the efficacy and side effects of autologous hematopoietic stem cell transplantation combined with CD19-CART for adult acute lymphoblastic leukemia, and to evaluate the safety and efficacy of this regimen in the treatment of acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with high-risk acute B-lymphoblastic leukemia
* Complete remission was achieved after induction chemotherapy, and autologous CD19-CAR-T was successfully prepared
* Eligible for autologous hematopoietic stem cell transplantation
* No major organ dysfunction

Exclusion Criteria:

* Combined with malignant tumors of other organs
* With a serious infection that is not under control
* Syphilis, AIDS, hepatitis B, hepatitis C, any one of them positive
* Patients who have had an allergic reaction to the drugs used in this study or similar drugs
* Other patients deemed unsuitable for inclusion by the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Relapse rate within 2 years | Time Frame: From autologous hematopoietic stem cell transplantation to 2 years after transplantation

SECONDARY OUTCOMES:
Non-relapse mortality | Time Frame: From autologous hematopoietic stem cell transplantation to 2 years after transplantation
Progression-free survival | Time Frame: From autologous hematopoietic stem cell transplantation to 2 years after transplantation
Overall survival rate | Time Frame: From autologous hematopoietic stem cell transplantation to 2 years after transplantation
Incidence of infection | Time Frame: From autologous hematopoietic stem cell transplantation to 2 years after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- NO.288 Nanjing Road，Heping District，Tianjin, Tianjin,, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Haven't thought it through yet